CLINICAL TRIAL: NCT04330326
Title: A Phase 2, Randomised, Placebo Controlled Study to Evaluate the Efficacy, Tolerability and Safety of Metabolic Cofactor Supplementation in Obese Subjects With Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Metabolic Cofactor Supplementation in Obese Patients With Non-Alcoholic Fatty Liver Disease
Acronym: NAFLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ScandiBio Therapeutics AB (Industry)
Collaborators: Koç University (Other); Koç University Hospital (Unknown); Göteborg University (Other); Sahlgrenska University Hospital (Other); KTH Royal Institute of Technology (Other); University of Helsinki (Other); Helsinki University Central Hospital (Other); Monitor CRO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 309
Record Dates: First submitted 2020-03-27; First posted 2020-04-01 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Sorbitol

STUDY DESIGN:
Intervention Model Description: A total of 45 overweight or obese patients with NAFLD will be randomized on a 2:1 basis to the cofactor mixture or placebo.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Subjects in active treatment will receive dietary supplementation with N-acetylcysteine, L-carnitine tartrate, nicotinamide riboside, and serine, administered as a mixture.
  Interventions: Drug: Metabolic Cofactor Supplementation
- Placebo Arm (Placebo Comparator): Subjects will take a mixture of placebo as powder dissolved in water by mouth.
  Interventions: Drug: Sorbitol

INTERVENTIONS:
Drug: Metabolic Cofactor Supplementation — Subjects in active treatment will receive dietary supplementation with N-acetylcysteine, L-carnitine tartrate, nicotinamide riboside, and serine, administered as a mixture. Half dosage of the co-factors will be given for two weeks (one dose taken just after dinner), and full dosage for 8 weeks (two equal doses taken just after breakfast and dinner).
  Arms: Treatment Arm
Drug: Sorbitol — As placebo, sorbitol (5 g) flavored with strawberry aroma and coloring agent will be given. Sorbitol is widely used due to its solubility in water. It's approved by the U.S. Food and Drug Administration (FDA).
  Arms: Placebo Arm

SUMMARY:
This short-term, randomized, placebo-controlled, investigator-initiated trial aims to establish metabolic improvements in NAFLD subjects by dietary supplementation with cofactors N-acetylcysteine, L-carnitine tartrate, nicotinamide riboside and serine. Concomitant use of pivotal metabolic cofactors via simultaneous dietary supplementation will stimulate three different pathways to enhance hepatic β-oxidation and this study's hypothesis is that this will result in decreased amount of fat in the liver.

DETAILED DESCRIPTION:
In this study, investigators aim to lower liver fat content in obese patients with NAFLD by increasing the hepatic levels of pivotal metabolic cofactors via simultaneous dietary supplementation of serine, L-carnitine, N-acetylcysteine (NAC) and nicotinamide riboside (NR).

The study is based on a three-step strategy to increase the amount of fat oxidization in liver: (1) First, the investigators will include L-carnitine to enhance the transport of fatty acids across the mitochondrial membrane (by forming a long chain acetylcarnitine ester and being transported by carnitine palmitoyltransferase (CPT) I and CPT II). Carnitine also plays a role in stabilizing coenzyme A (CoA) and acetyl-CoA levels through the ability to receive or give an acetyl group. (2) Second, the investigators will include nicotinamide riboside, precursor of nicotinamide adenine dinucleotide (NAD+) to boost the level of hepatic β-oxidation of fatty acids in mitochondria. Decreased electron transport chain function combined with impaired rates of fatty acid β-oxidation leads to the accumulation of incomplete products of β-oxidation, which combined with increased levels of reactive oxygen species (ROS) contribute to insulin resistance. Furthermore, as L-carnitine, nicotinamide

riboside stimulate the transfer of fatty acids from cytosol to mitochondria.(3) Finally, they will include the two glutathione precursors serine and N-acetylcysteine to increase glutathione levels in the hepatocytes. Increased glutathione levels will also protect against free radical-mediated oxidative stress generated by the increased β-oxidation of fatty acids in mitochondria.

Previous studies showed that each agent is able to decrease liver fat amount separately and a proof-of-concept study using serine supplementation, and a phase I study using this three-step approach resulted in a significant decrease in plasma metabolites associated with liver fat without significant side effect. Concomitant use of pivotal metabolic cofactors via simultaneous dietary supplementation will stimulate three different pathways to enhance hepatic β-oxidation. The novel design with this study is to give the L-carnitine, NR, serine and NAC as a cocktail. Based on investigators' hypothesis is that this will result in decreased amount of fat in the liver.

The study population will consist of 45 male and female adult overweight and obese subjects diagnosed with NAFLD. Eligible subjects must have signed an informed consent, meet all inclusion criteria and have none of the exclusion criteria. Patients will be randomized on a 2:1 basis to the cofactor mixture or placebo.

The subjects will take a mixture of cofactors or matching placebo as powder dissolved in water by mouth. Subjects in active treatment will receive dietary supplementation with N-acetylcysteine, L-carnitine tartrate, nicotinamide riboside, and serine, administered as a mixture. Half dosage of the co-factors will be given for two weeks (one dose taken just after dinner), and full dosage for 8 weeks (two equal doses taken just after breakfast and dinner). Patients who can tolerate the study agents will start to take half dose of co-factors supplementation (i.e., 1 dosage daily just after dinner) for two weeks.

The active treatment duration will be 10 weeks for each subject and the total study duration is estimated as 14 months. The study comprises seven clinical visits; (1) pre-screening visit, (2) screening visit, (2) randomization visit, (3) post-treatment visit (day 14); (4) post-treatment visit (day 28); (5) post-treatment visit (day 42) and (4) end of treatment visit (day 70). At visit 1 informed consent will be signed, all procedures including clinical and physical examination, assessment of inclusion and exclusion criteria, genetic analysis and transient elastography will be done. At visit 2 and visit 7, all procedures including review of 3-day diet records, clinical and physical examination; body composition analysis with Bioelectrical Impedance Analysis (BIA), ECG evaluation, blood, urine and stool sampling for routine laboratory tests, lipidomics, metabolomics and gut microbiota analysis and magnetic resonance imaging and MR spectroscopy will be carried out. At visit 3, eligible study subjects will be randomized to active therapy or placebo groups and study agents will be dispensed as half-of therapy. At visit 4, and 6, clinical and physical examination, ECG evaluation, blood, urine and stool sampling for routine laboratory tests, lipidomics, metabolomics and gut microbiota analysis, magnetic resonance imaging and MR spectroscopy and initiation of full dose therapy (i.e. taking cocktails two times just after breakfast and dinner) will be realized. At visit 5, visit 4 and 6 will be repeated excluding magnetic resonance imaging and MR spectroscopy. After the visit 7, participants will stop taking study agents.

A subject will be considered as having completed the study if he/she has completed all assessments at the End of Treatment Visit (Visit 7) and has been followed up until 10 weeks after initiation of the study drugs.

Statistics for the primary outcome parameter will be tested by Mann-Whitney U test or t-test depending on the results of normality test. For the secondary and third outcome parameters one-way repeated measures ANOVA will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (18-70 years old)
* Body mass index >27kg/m2
* Triglyceride levels ≤354 mg/dl and LDL chol ≤175 mg/dl
* No history of medication use for hepatic steatosis
* Increased liver fat (>5.5%)

Exclusion Criteria:

* Inability or unwillingness to give written informed consent
* Systolic blood pressure >160 mm Hg and/or diastolic blood pressure > 105 mm Hg
* Type 1 or type 2 diabetes
* Chronic liver disease other than NAFLD (i.e. chronic infection with hepatitis C virus [HCV] or hepatitis B virus [HBV], autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson s disease, alpha-1 antitrypsin deficiency).
* Previous gastric or small bowel surgery
* Active gastric ulcer
* Inflammatory bowel disease
* ALT or AST >3× ULN (upper limit of normal)
* Detection of cirrhosis by transient elastography or other imaging modalities
* Diarrhea (defined as more than 2 stool per day) within 7 days before enrollment
* Chronic kidney disease with an estimated glomerular filtration rate <60 ml/min/1.73m2
* Significant cardiovascular co-morbidity (i.e. heart failure, documented coronary artery disease, valvular heart disease)
* Patients with active bronchial asthma
* Patients with phenylketonuria (contraindicated for NAC)
* Patients with histamine intolerance
* Clinically significant TSH level outside the normal range (0.04-6 mU/L)
* Known allergy for substances used in the study
* Concomitant medication use:

  1. Lipid-lowering drugs within 3 months
  2. Oral antidiabetics given for insulin resistance of obesity (metformin, liraglutide etc.) within 3 months
  3. Thiazide diuretics with a dose >25 mg/d
  4. Postmenopausal estrogen therapy
  5. Any medication acting on nuclear hormone receptors or inducing Cytochromes P450 (CYPs)
  6. Self-administration of dietary supplements such as any vitamins, omega-3 products, or plant stanol/sterol products within 1 month
  7. Treatment with medications known to cause fatty liver disease such as atypical neuroleptics, tetracycline, methotrexate or tamoxifen
  8. Use of an antimicrobial agent in the 4 weeks preceding randomization
* Active smokers consuming >10 cigarettes/day
* Alcohol consumption over 192 grams for men and 128 grams for women per week
* Patients considered as inappropriate for this study for any reason (patients unable to undergo MRI study, noncompliance etc.)
* Subjects with Patatin-like phospholipase domain-containing protein 3( PNPLA3) I148M (homozygous for I148M)
* Women who are pregnant, are planning pregnancy, or who are breast-feeding
* Women of childbearing potential not protected by effective birth control method
* Active participation in another clinical study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Spectroscopy (MRS) Measurement | 2 weeks, 6 weeks and 10 weeks
  The change in liver fat content as well as subcutaneous abdominal and intra-abdominal fat content between the placebo and cofactor treatment arms in NAFLD patients from baseline to 2 weeks, 6 weeks and 10 weeks.

SECONDARY OUTCOMES:
Change in body weight from baseline | 10 weeks
  Body weight will be measured at every visit to evaluate safety of metabolic cofactor supplementation.
ECG Measurement | 10 weeks
  Change in heart rate will be measured at every visit to evaluate safety of metabolic cofactor supplementation.
Change in Blood Pressure from baseline | 10 weeks
  Systolic and Diastolic Blood Pressure will be measured at every visit to evaluate safety of metabolic cofactor supplementation.
Change in waist and hip circumference from baseline | 10 weeks
  Waist and hip circumference will be measured at every visit to evaluate safety of metabolic cofactor supplementation.
Change of complete blood count (number of blood cells) from baseline | 10 weeks
  Complete blood count includes number of blood cells. Complete blood count test will be performed to measure possible toxic effects of the metabolic cofactor supplementation on hematological system.
Change of complete blood count (hemoglobin) from baseline | 10 weeks
  Complete blood count includes concentration of hemoglobin. Complete blood count test will be performed to measure possible toxic effects of the metabolic cofactor supplementation on hematological system.
Changes in kidney function tests (creatinine, urea, uric acid) from baseline | 10 weeks
  Kidney function tests (creatinine, urea, uric acid) will be performed to measure possible toxic effects of the metabolic cofactor supplementation on kidney function.
Changes in kidney function tests (sodium, potassium) from baseline | 10 weeks
  Kidney function tests (sodium, potassium) will be performed to measure possible toxic effects of the metabolic cofactor supplementation on kidney function.
Changes in liver function tests [Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Gamma-glutamyl transferase (GGT), Alkaline phosphatase (ALP)] from baseline | 10 weeks
  Liver function tests (ALT, AST, GGT, ALP) will be performed to measure possible toxic effects of the metabolic cofactor supplementation on liver function.
Changes in liver function tests (Total Bilirubin, and Albumin) from baseline | 10 weeks
  Liver function tests (Total Bilirubin, Albumin) will be performed to measure possible toxic effects of the metabolic cofactor supplementation on liver function.
Changes in creatinine kinase (CK) level from baseline | 10 weeks
  Creatinine kinase (CK) level will be evaluated to measure possible toxic effects of the metabolic cofactor supplementation.
Changes in blood lipid levels (total cholesterol (TC), triglyceride (TG), low density lipoprotein (LDL-C), high density lipoprotein (HDL-C)) from baseline | 2 weeks, 6 weeks and 10 weeks
  Blood lipid levels (total cholesterol (TC), triglyceride (TG), low density lipoprotein (LDL-C), high density lipoprotein (HDL-C)) will be evaluated to measure possible toxic effects of the metabolic cofactor supplementation.
Changes in blood glucose levels from baseline | 10 weeks
  Blood glucose levels will be evaluated to measure possible toxic effects of the metabolic cofactor supplementation.
Change in blood insulin level from baseline | 10 weeks
  Blood insulin level will be evaluated to measure possible toxic effects of the metabolic cofactor supplementation.
Change in thyroid-stimulating hormone (TSH) level from baseline | 10 weeks
  Thyroid-stimulating hormone (TSH) level will be evaluated to measure possible toxic effects of the metabolic cofactor supplementation.
Microbiota analysis | 2 weeks, 6 weeks and 10 weeks
  The change in gut microbiota between the placebo and the treatment arms in NAFLD patients. Feces and saliva samples will be collected to assess changes in gut microbiota. Instructions on specimen collection will be given during the first visit. Microbiota will be assessed using shot-gun metagenomic techniques.
Monitoring of adverse events | 10 weeks
  This process aiming to monitoring of adverse events of metabolic cofactor supplementation. Adverse events and serious adverse events will be monitored continuously and all adverse events that occur at any time during the study will be reported in Case Report Forms. Any symptoms of intestinal discomfort or other side effects will be carefully recorded and all study subjects will be informed to contact (by phone or text message) the investigators immediately if they experience any symptoms of discomfort or any side effects during the intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Koç University Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Zeybel M, Altay O, Arif M, Li X, Yang H, Fredolini C, Akyildiz M, Saglam B, Gonenli MG, Ural D, Kim W, Schwenk JM, Zhang C, Shoaie S, Nielsen J, Uhlen M, Boren J, Mardinoglu A. Combined metabolic activators therapy ameliorates liver fat in nonalcoholic fatty liver disease patients. Mol Syst Biol. 2021 Oct;17(10):e10459. doi: 10.15252/msb.202110459. PMID 34694070